CLINICAL TRIAL: NCT06784661
Title: Immediate Effects of Lipid-Based Artificial Tears (Mineral Oil and Hydroxypropyl Guar) and Non-Lipid Artificial Tears (Hydroxypropyl Guar) on Corneal Aberrations in Healthy Individuals
Brief Title: Immediate Effects of Lipid-Based and Non-Lipid Artificial Tears on Corneal Aberrations
Acronym: ILEACT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, José-María Sánchez-González, Optometry Doctor, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USeville_2025_01
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Aberration, Corneal Wavefront
Keywords: Corneal aberrations; Aberrations; Wavefront
MeSH Terms: conditions — Corneal Wavefront Aberration

STUDY DESIGN:
Intervention Model Description: This parallel design allows for comparison of the effects of each formulation across two distinct groups. Each participant will receive a single application of their assigned formulation, and the effects will be measured uniformly at specific time points.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and outcomes assessors will not know which formulation is being administered. Identical containers and consistent procedures will ensure masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lipid-Based Artificial Tear Formulation (Experimental): Participants in this arm will receive a single drop of a lipid-based artificial tear formulation containing mineral oil and hydroxypropyl guar in each eye. The intervention is designed to enhance the lipid layer of the tear film and will be evaluated for its immediate effects on corneal aberrations 15 minutes post-instillation.
  Interventions: Drug: Lipid-Based Artificial Tear
- Non-Lipid Artificial Tear Formulation (Experimental): Participants in this arm will receive a single drop of a non-lipid artificial tear formulation containing hydroxypropyl guar in each eye. The intervention aims to improve aqueous layer stability and will be assessed for its immediate effects on corneal aberrations 15 minutes post-instillation.
  Interventions: Drug: Non-Lipid Artificial Tear

INTERVENTIONS:
Drug: Lipid-Based Artificial Tear — This intervention consists of a lipid-based artificial tear formulation containing mineral oil and hydroxypropyl guar. It is designed to enhance the tear film's lipid layer and improve ocular surface stability. Participants in this group will receive a single drop in each eye, and corneal aberrations will be measured at baseline and 15 minutes after instillation.
  Arms: Lipid-Based Artificial Tear Formulation
Drug: Non-Lipid Artificial Tear — This intervention consists of a non-lipid artificial tear formulation containing hydroxypropyl guar. It is intended to stabilize the aqueous layer of the tear film and maintain optical quality. Participants in this group will receive a single drop in each eye, and corneal aberrations will be measured at baseline and 15 minutes after instillation.
  Arms: Non-Lipid Artificial Tear Formulation

SUMMARY:
This study evaluates the immediate effects of two types of artificial tear formulations on corneal aberrations in a healthy population. The interventions include a lipid-based formulation containing mineral oil and hydroxypropyl guar, and a non-lipid formulation containing hydroxypropyl guar alone. Participants will receive a single instillation of each formulation in separate eyes, with measurements of corneal aberrations taken before and 15 minutes after instillation. The study aims to compare the optical changes induced by these formulations and assess their impact on the ocular surface quality.

DETAILED DESCRIPTION:
This study explores the immediate effects of two types of artificial tear formulations on corneal aberrations in healthy individuals. The primary aim is to evaluate how a lipid-based formulation containing mineral oil and hydroxypropyl guar and a non-lipid formulation containing hydroxypropyl guar alone influence optical quality shortly after instillation. The results of this research will contribute to a better understanding of how these formulations interact with the ocular surface to enhance or alter corneal optical properties.

The study will involve healthy participants aged 18 to 35 years, with no prior history of ocular surface disease, refractive surgery, or contact lens use. All participants will undergo a baseline assessment of corneal aberrations before any intervention. Each individual will then receive a single drop of the lipid-based formulation in one eye and the non-lipid formulation in the other eye. This approach allows for direct comparison between the two interventions within the same participant. Measurements of corneal aberrations will be taken 15 minutes after instillation to capture the immediate effects of each formulation on optical quality.

The study is designed as a randomized, participant-masked clinical trial to ensure unbiased results. By measuring higher-order aberrations (HOAs) with wavefront aberrometry, the research will assess how these artificial tears affect the ocular surface's optical properties. This will provide valuable insights into their potential to stabilize the tear film and enhance visual performance. The trial follows ethical guidelines and has been approved by the appropriate Institutional Review Board.

This research is important for advancing knowledge about artificial tear formulations and their role in managing ocular surface conditions. Although both formulations are commonly used in clinical practice, their specific effects on corneal aberrations immediately after application have not been thoroughly studied in a healthy population. The findings from this study will help inform healthcare providers and patients about the optical benefits and limitations of these widely used artificial tear formulations.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals aged 18 to 35 years. No prior history of ocular surface disease, refractive surgery, or contact lens wear.

Corrected visual acuity of 20/20 or better. Ability to provide informed consent. Willingness to comply with study procedures, including instillation of artificial tears and follow-up measurements.

Exclusion Criteria:

History of any ocular surgery or trauma within the past six months. Use of any systemic or topical medications that may affect ocular surface stability or tear film.

Any active or chronic ocular infection, inflammation, or other pathology. Known hypersensitivity or allergy to any components of the artificial tears. Pregnancy or breastfeeding. Participation in another clinical trial within the last 30 days.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Corneal Higher-Order Aberrations (HOAs) | Baseline to 15 minutes post-instillation
  The primary outcome is the change in corneal higher-order aberrations (measured as RMS values) using wavefront aberrometry. Measurements will assess the optical impact of the lipid-based and non-lipid artificial tear formulations on the ocular surface.

SECONDARY OUTCOMES:
Stabilization of Tear Film | Baseline to 15 minutes post-instillation
  This outcome evaluates the qualitative stabilization of the tear film post-instillation of the artificial tear formulations. Observations will include tear film uniformity and potential disruptions measured indirectly through aberrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- ISEC Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to privacy and confidentiality concerns. The data collected in this study will be used solely for the purposes outlined in the research protocol and will remain confidential according to applicable data protection regulations. Aggregate data and study results will be shared in peer-reviewed publications and presentations, but individual-level data will not be made publicly available.

REFERENCES:
- [Background] Yildirim Y, Ozsaygili C, Kucuk B. The short term effect of trehalose and different doses of sodium hyaluronate on anterior corneal aberrations in dry eye patients. Cutan Ocul Toxicol. 2021 Mar;40(1):14-20. doi: 10.1080/15569527.2020.1861001. Epub 2020 Dec 21. PMID 33342322
- [Background] Lee H, Kim SM, Choi S, Seo KY, Kim EK, Kim TI. Effect of diquafosol three per cent ophthalmic solution on tear film and corneal aberrations after cataract surgery. Clin Exp Optom. 2017 Nov;100(6):590-594. doi: 10.1111/cxo.12521. Epub 2017 Feb 21. PMID 28222481
- [Background] Mihaltz K, Faschinger EM, Vecsei-Marlovits PV. Effects of Lipid- Versus Sodium Hyaluronate-Containing Eye Drops on Optical Quality and Ocular Surface Parameters as a Function of the Meibomian Gland Dropout Rate. Cornea. 2018 Jul;37(7):886-892. doi: 10.1097/ICO.0000000000001523. PMID 29377842
- [Background] Lekhanont K, Chuckpaiwong V, Vongthongsri A, Sangiampornpanit T. Effects of sodium hyaluronate on wavefront aberrations in dry eye patients. Optom Vis Sci. 2014 Jan;91(1):39-46. doi: 10.1097/OPX.0000000000000101. PMID 24366433
- [Background] Habbe KJ, Frings A, Saad A, Geerling G. The influence of a mineral oil cationic nanoemulsion or perfluorohexyloctane on the tear film lipid layer and higher order aberrations. PLoS One. 2023 Jan 18;18(1):e0279977. doi: 10.1371/journal.pone.0279977. eCollection 2023. PMID 36652431
- [Background] Saad A, Frings A. Influence of perfluorohexyloctane (Evotears(R)) on higher order aberrations. Int Ophthalmol. 2023 Dec;43(12):5025-5030. doi: 10.1007/s10792-023-02905-w. Epub 2023 Oct 21. PMID 37864619
- [Background] Carpena-Torres C, Pastrana C, Rodriguez-Pomar C, Serramito M, Batres L, Carracedo G. Changes in visual quality with soft contact lenses after the instillation of hyaluronic acid eye drops. Cont Lens Anterior Eye. 2021 Dec;44(6):101471. doi: 10.1016/j.clae.2021.101471. Epub 2021 May 26. PMID 34049809
- [Derived] Sanchez-Gonzalez JM, Sanchez-Gonzalez MC, De-Hita-Cantalejo C, Nascimento H, Martinez-Perez C. Immediate Impact of Artificial Tear Composition on Optical Aberrations: A Comparative Study of Lipid and Non-Lipid Hydroxypropyl Guar Formulations. Ophthalmol Ther. 2025 Sep;14(9):2165-2178. doi: 10.1007/s40123-025-01205-z. Epub 2025 Jul 17. PMID 40676409